CLINICAL TRIAL: NCT01101204
Title: Effects of High and Low Doses of Metformin, Fenofibrate and Simvastatin, Administered Together and in Sequence With Lifestyle Intervention on Lipid Profile, Glucose Metabolism, Low-grade Inflammation and Hemostasis in Patient's Blood Plasma in Type 2 Diabetic Patients With Serious Mixed Dyslipidemia
Brief Title: The Effects of Hypolipemic and Antidiabetic Treatment on Cytokines
Acronym: MSF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Bogusław Okopień, MD PhD, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MSF
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes; Dyslipidemia; Inflammation; Cytokines
MeSH Terms: conditions — Diabetes Mellitus; Dyslipidemias; Inflammation | interventions — Metformin; Simvastatin; Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- M1000 S10 F100 (Active Comparator): metformin 1000mg, fenofibrate 100mg and simvastatin 10mg
  Interventions: Drug: Metformin 1000mg, simvastatin 10mg and fenofibrate 100mg
- M1000 S10 F267 (Active Comparator): metformin 1000mg, fenofibrate 267mg and simvastatin 10mg
  Interventions: Drug: Metformin 1000mg, simvastatin 10mg and fenofibrate 100mg
- M1000 S40 F100 (Active Comparator): metformin 1000mg, fenofibrate 100mg and simvastatin 40mg
  Interventions: Drug: Metformin 1000mg, simvastatin 10mg and fenofibrate 100mg
- M1000 S40 F267 (Active Comparator): metformin 1000mg, fenofibrate 267mg and simvastatin 40mg
  Interventions: Drug: Metformin 1000mg, simvastatin 10mg and fenofibrate 100mg
- M2500 S10 F100 (Active Comparator): metformin 2500mg, fenofibrate 100mg and simvastatin 10mg
  Interventions: Drug: Metformin 1000mg, simvastatin 10mg and fenofibrate 100mg
- M2500 S10 F267 (Active Comparator): metformin 2500mg, fenofibrate 267mg and simvastatin 10mg
  Interventions: Drug: Metformin 1000mg, simvastatin 10mg and fenofibrate 100mg
- M2500 S40 F267 (Active Comparator): metformin 2500mg, fenofibrate 267mg and simvastatin 40mg
  Interventions: Drug: Metformin 1000mg, simvastatin 10mg and fenofibrate 100mg
- M2500 S40 F100 (Active Comparator): metformin 2500mg, fenofibrate 100mg and simvastatin 40mg
  Interventions: Drug: Metformin 1000mg, simvastatin 10mg and fenofibrate 100mg
- Therapeutic Lifestyle Change (Placebo Comparator): Only therapeutic lifestyle change
  Interventions: Drug: Metformin 1000mg, simvastatin 10mg and fenofibrate 100mg

INTERVENTIONS:
Drug: Metformin 1000mg, simvastatin 10mg and fenofibrate 100mg — Patient will take three pill consisting of metformin 1000mg, simvastatin 10mg and fenofibrate 100mg.

SUMMARY:
The study is planned to show whether combined hypolipemic and antidiabetic therapy with various daily dosages influence the fasting plasma glucose, insulin sensitivity and proinflammatory cytokines in diabetic and dyslipidemic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age (35-64yr)
* Primary hyperlipidemia (Total cholesterol >200mg/dl, Triglycerides >150mg/dl)
* Type 2 Diabetes
* For women:
* Menopause (>12 months)
* Post hysterectomy
* Mechanical contraception
* Obtained informed consent

Exclusion Criteria:

* Secondary hyperlipidemia
* Morbid obesity (BMI>40kg/m2)
* Alcohol or drug abuse
* Acute or chronic inflammation
* Congestive Heart Failure (NYHA III or IV)
* Unstable Ischaemic Heart Disease
* Moderate or severe hypertension
* Cancer in less than 5 years
* Chronic kidney disease (stage III-V)
* Liver failure
* Oral contraception
* Not compliant patient
* Laboratory results:
* alanine transferase (>3xULN)
* creatine kinase (>5xULN)
* haemoglobin (<10/dl)
* PLT (<100G/l)
* WBC (<3,5G/l or >10G/l)

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Antiinflammatory effects of combined antidiabetic and hypolipemic treatment | 30 days
  As inflammatory effects we measure the difference in serum concentration before and after the treatment of the following proinflammatory cytokines:
  1. Interleukin 1
  2. TNF alpha
  3. Interleukin 6
  4. Interleukin 10
  5. hsCRP

SECONDARY OUTCOMES:
Insulin sensitivity | 30 days
  Assesed by HOMA (Homeostatic Model of Assessment)
Coagulation parameters | 30 days
  Assessed using:
  1. Fibrinogen
  2. PAI-1

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Katowice, Katowice, Poland